CLINICAL TRIAL: NCT07311954
Title: Development and Validation of a cCTA and Biomarker Based Risk Model for Coronary Revascularization in Elderly Patients With Coronary Artery Disease
Status: Not yet recruiting | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Collaborators: Central China Fuwai Hospital of Zhengzhou University (Other); Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-2970
Record Dates: First submitted 2025-12-17; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Coronary Artery Disease; Elderly (Aged >70)
Keywords: coronary computed tomography angiography; frailty; biomarker
MeSH Terms: conditions — Coronary Artery Disease; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Model Development and Validation Cohort
  Interventions: Other: No Intervention: Observational Cohort

INTERVENTIONS:
Other: No Intervention: Observational Cohort — No intervention will be conducted.

SUMMARY:
This study is a prospective multi-center observational cohort involving elderly patients (≥70 years old) with multi-vessel coronary disease identified by coronary computed tomography angiography (cCTA) and scheduled for invasive coronary angiography. Data collection about cCTA, frailty and biomarkers and two-year follow-up will be conducted to develop and validate a risk model of coronary revascularization.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 70 years.
2. Multivessel coronary artery disease identified on coronary computed tomography angiography (CCTA), defined as ≥50% stenosis in at least two of the three major epicardial coronary arteries.
3. Scheduled to undergo invasive coronary angiography as part of standard clinical care.
4. Able to provide informed consent, or consent provided by a legally authorized representative.

Exclusion Criteria:

1. Previous coronary revascularization, including percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABG).
2. Acute myocardial infarction at admission, according to electrocardiographic findings and elevated cardiac biomarkers consistent with acute MI.
3. Poor-quality CCTA images that prevent accurate assessment of coronary plaque characteristics or stenosis severity.
4. Refusal or inability to participate in the study or to provide informed consent.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients aged 70 years and older with multivessel coronary artery disease identified by coronary CT angiography and scheduled to undergo invasive coronary angiography at participating centers.
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Area Under the Receiver Operating Characteristic Curve (AUC) for Risk Model Performance | At completion of 2-year follow-up
  AUC evaluates the model's discrimination performance in predicting MACCEs at 24 months.

SECONDARY OUTCOMES:
Sensitivity of the Prediction Model | At completion of 2-year follow-up
  The proportion of participants who actually experienced MACCEs (Major Adverse Cardiac and Cerebral Events) that were correctly identified by the prediction model as high risk.
Specificity of the Prediction Model | At completion of 2-year follow-up
  The proportion of participants who did not experience MACCEs that were correctly identified by the prediction model as low risk.
Positive Predictive Value (PPV) | At completion of 2-year follow-up
  The probability that subjects identified by the model as high risk truly experienced the adverse events (MACCEs).
Negative Predictive Value (NPV) | At completion of 2-year follow-up
  The probability that subjects identified by the model as low risk truly did not experience the adverse events.
Hosmer-Lemeshow Goodness-of-Fit Statistic | At completion of 2-year follow-up
  A statistical test to assess the calibration of the model. It evaluates whether the observed event rates match the expected event rates in subgroups of the model population. A non-significant p-value indicates good fit.
Calibration Slope | At completion of 2-year follow-up
  Assessment of the agreement between observed outcomes and predicted risks. A slope (beta) of 1 indicates ideal calibration.
Decision Curve Analysis (DCA) | At completion of 2-year follow-up
  Evaluation of clinical net benefit across a range of threshold probabilities.

IPD SHARING:
Plan to Share IPD: No